CLINICAL TRIAL: NCT06311175
Title: Mentoring in Mobile Health (mHealth) and Social Networking Interventions for Cardiovascular Disease Risk Reduction: Intervention Phase
Brief Title: Diet Tracking Prescriptions for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Sherry Pagoto, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H20-0114
Record Dates: First submitted 2024-01-03; First posted 2024-03-15 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three intervention groups in parallel for the duration of the study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Diet Tracking Prescription (Active Comparator): This group will be asked to track their diet using a commercial mobile application every day for the 8 week digital weight loss intervention.
  Interventions: Behavioral: Dietary Tracking Prescription
- 66% Tracking Prescription (Experimental): This group will be asked to track their diet for 2 weeks, then they will get a 1 week break, track for 2 more weeks and then get a 1 week break, and then track for 2 weeks during the 8 week digital weight loss intervention.
  Interventions: Behavioral: Dietary Tracking Prescription
- 50% Tracking Prescription (Experimental): This group will be asked to track their diet every other week during the 8 week digital weight loss intervention.
  Interventions: Behavioral: Dietary Tracking Prescription

INTERVENTIONS:
Behavioral: Dietary Tracking Prescription — Dietary tracking prescriptions to follow during a digital weight loss intervention.

SUMMARY:
Lifestyle interventions are effective at producing modest weight loss. One of the strongest predictors of weight loss is food tracking, which involves logging all food and beverage consumed each day in an effort to stay within a daily calorie goal. Standard lifestyle interventions prescribe daily food tracking for the length of the program which can range from 3-24 months. This can be a taxing prescription that is not feasible to do long term for many people. The purpose of this pilot feasibility randomized trial is to test the feasibility of 3 tracking prescriptions during an 8 week digital weight loss intervention: 1) tracking daily, 2) tracking two weeks on and one week off, 3) tracking every other week. Feasibility is defined as tracking prescription compliance, burden, acceptability, and perceived efficacy, and tracking self-efficacy. Diet tracking will be evaluated one month after the intervention ends so that groups can be compared on diet tracking maintenance.

DETAILED DESCRIPTION:
The investigators propose a pilot randomized feasibility trial in which they will randomize 108 people to 3 remotely-delivered weight loss intervention groups that vary based on their diet tracking prescription. The primary outcome will be feasibility, acceptability, and perceived efficacy of the "lighter" tracking prescriptions. Each group will have 36 participants and the intervention will last 8 weeks. They will do assessments at baseline, 8 weeks, and 12 weeks. The 8 week assessment will include weight, diet tracking records, and a survey on acceptability. The 12 week assessment will evaluate weight and diet tracking in the month following the intervention which will allow them to explore diet tracking persistence in that time period. All three intervention groups will receive the same remotely delivered lifestyle intervention, but will vary based on three different tracking prescriptions: 1) Standard Diet Tracking Prescription: This group will be asked to track their diet every day for 8 weeks.

2) 66% Tracking Prescription. This group will be asked to track for 2 weeks, then they will get a 1 week break, track for 2 more weeks and then get a 1 week break, and then track for 2 weeks. 3) 50% Tracking Prescription. This group will be asked to track every other week which would result in 4 weeks of tracking and 4 weeks off of tracking. The primary outcome of this trial is feasibility as defined as: 1) compliance with the tracking prescription (i.e., % of prescribed days with complete tracking, % tracking in week 8) 2) burden of tracking prescription (e.g., time consuming, hard to remember) 3) acceptability of tracking prescription (e.g., ease, plans to continue the prescription) 4) perceived efficacy of tracking prescription (e.g., "tracking this often is enough to help me lose weight"). 5) self-efficacy of diet tracking (e.g., "I feel confident I could continue this tracking prescription for the next 3 months"). 6) number of diet tracking days in the subsequent month. Percent weight loss at 8 and 12 weeks in each group will be exploratory outcomes and presented descriptively as this pilot is not powered to establish efficacy. Feasibility hypotheses and/or benchmarks are as follows:

1. Tracking Adherence Hypothesis: Participants in groups 2 and 3 will have completed a significantly higher proportion of days of their total prescription than group 1. This will inform the future trial by demonstrating that adherence to the new prescriptions is higher than the standard prescription.
2. Tracking Persistence Hypothesis: Participants in groups 2 and 3 will have tracked significantly more days in week 8 (last week of intervention) than participants in group 1. This will inform the future trial by demonstrating that a higher proportion of participants receiving the new prescriptions will still be tracking at week 8 than participants in the standard prescription. This is evidence that the abbreviated tracking prescriptions may result in a longer term tracking than the standard prescription.
3. Tracking Burden Hypothesis: Participants in groups 2 and 3 will rate the burden of their tracking prescription significantly lower than participants in group 1. This will inform the future trial by demonstrating that the lighter tracking prescriptions will be viewed as less burdensome, which is further evidence that participants may be willing to track longer if they feel less burdened by the task.
4. Tracking Acceptability Hypothesis: Participants in groups 2 and 3 will rate the acceptability of their tracking prescription significantly higher than participants in group 1. This will inform the future trial by demonstrating that the lighter tracking prescriptions will be viewed as more acceptable, which is further evidence that participants may be willing to track longer if they feel the task is easier.
5. Perceived Efficacy Benchmark: At least 80% of participants in all groups will rate the perceived efficacy of their tracking prescription for weight loss to be high to very high. This will inform the future trial by demonstrating that the lighter tracking prescriptions are viewed by most as enough to result in weight loss. The investigators want to be careful that they do not lose faith in a lighter tracking prescription so they are testing two different light versions.
6. Self-Efficacy for Tracking Hypothesis: Participants in groups 2 and 3 will have higher self-efficacy for their diet tracking prescription compared to group 1 and group 3 will have higher self-efficacy than group 2. This will inform the future trial by demonstrating that participants given the lighter tracking prescriptions will have higher self-efficacy for diet tracking which may be another indication that they may be willing to track over a longer period of time compared to the standard tracking prescription.
7. Post-Intervention Tracking Adherence Benchmark: At least 80% of participants in groups 2 and 3 will match their diet tracking prescription in the subsequent month. This will inform the future trial by showing evidence for a high level of consistency for the lighter tracking prescriptions. If one of the two lighter prescriptions meets this benchmark, the investigators will select it for testing in the subsequent trial.
8. Post-Intervention Tracking Prescription Hypothesis: A significantly higher proportion of participants in groups 2 and 3 will have tracked in the final week of the subsequent month compared to participants in group 1. This will inform the future trial by providing evidence that the lighter tracking prescriptions will lead to longer term tracking than the standard condition where tracking goes down precipitously over 2-3 months.

Findings from this pilot randomized feasibility trial will be used to inform an efficacy trial comparing one or both "light" tracking prescriptions to the standard tracking prescription on weight loss at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-45 kg/m2
* Wi-Fi connectivity at home
* Logs into Facebook at least 5 days per week over the past 2 weeks
* Has "liked", posted, or replied on Facebook at least twice a week over the past month
* Able to participate in the study in English
* Interested in losing weight
* Lives in US

Exclusion Criteria:

* Pregnant/lactating or plans to become pregnant during study period
* Reports having bipolar disorder, substance abuse, psychosis, an eating disorder, or severe depression
* Had bariatric surgery or plans to have surgery during the study
* Currently taking medication affecting weight
* Has lost ≥5% of weight in past 3 months
* Is participating or intends to participate in another weight loss program during the study
* Chronic pain that interferes with the ability to exercise
* Type 1 Diabetes
* Type 2 Diabetes
* Unable to make dietary changes or increase physical activity
* Unable to walk ¼ mile unaided without stopping
* Currently smokes or vapes nicotine twice a week or more
* Has a digestive disorder/condition that precludes dietary changes
* Meets criteria for severe depression on the Patient Health Questionnaire-8 (score of >19)
* Does not currently own a smartphone
* Participated in previous weight loss studies under the PI
* Unable to attend the orientation webinar
* Had major surgery in past 6 months and have not been cleared by their doctor to resume physical activity and diet changes
* Plans to have major surgery in the next 6-months
* Has an implanted cardiac defibrillator or pacemaker
* Did not complete screening and on-board processes of study (screening survey, webinar, e-consent, baseline survey, app set-up, scale set-up, etc.)
* Prisoner; or
* Unable to provide consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Compliance with diet tracking prescription | 8 weeks
  percent of prescribed days with complete tracking
Persistence with diet tracking prescription | 8 weeks
  percent of days of complete tracking in week 8
Burden of tracking prescription | 8 weeks
  Total score of three items: 5 point Likert scale ratings of how time consuming, hard to remember, and stressful the prescription was to follow. Minimum score =0, maximum score =12. Higher scores indicate higher burden
Acceptability of tracking prescription | 8 weeks
  Total score of three items: 5 point Likert scale ratings of how easy the tracking prescription is, how much they like it, and their plans to continue the tracking prescription. Minimum score =0, maximum score =12. Higher scores indicate higher acceptability.
Perceived efficacy of tracking prescription | 8 weeks
  Total score of how much they agree with 3 items on a 5 point Likert scale: tracking this often is enough to help me lose weight, tracking this often is enough to help me eat a healthier diet, and tracking this often is enough to keep me exercising. Minimum score =0, maximum score =12. Higher scores indicate higher perceived efficacy.
Self-efficacy of diet tracking | 8 weeks
  Total score of how much they agree with 3 items on a 5 point Likert scale: "I feel confident I could continue this tracking prescription for the next month." "I feel confident I could continue this tracking prescription for 3 months." "I feel confident I can continue this tracking prescription for 6 months." Minimum score =0, maximum score =12. Higher scores indicate higher self-efficacy.

SECONDARY OUTCOMES:
Diet Tracking One Month Post-Intervention | 12 weeks
  Number of diet tracking days in the subsequent month

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Pagoto, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT06311175/Prot_000.pdf
  • Informed Consent Form (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT06311175/ICF_001.pdf